CLINICAL TRIAL: NCT04708808
Title: The Efficacy of Music as an Adjunct Analgesic in Reducing Pain and Anxiety During Ultrasound-guided Manual Vacuum Aspiration (USG-MVA): A Randomized Controlled Trial
Brief Title: The Effect of Music Therapy Under Ultrasound Guided Manual Vacuum Aspiration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.0503
Record Dates: First submitted 2020-09-18; First posted 2021-01-14 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: First Trimester Abortion; Surgical Abortion; Music Intervention; Local Anesthesia; Pain
Keywords: music; termination of pregnancy; suction curettage; evacuation of gestational product; anxiety; abortion; pain; surgical abortion; aspiration abortion
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: First trimester miscarriage case undergo the manual vaccum procedure.
Masking Description: For those who consented to the study, they will be randomly assigned to receive music therapy or no according to a computer generated random number series. Each number will be placed in an opaque envelope labelled serially: (i) intervention group: routine care plus music given via headphone (ii) control group- routine care with no music or headphones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MVA case undergone music therapy (Experimental): case undergone manual vacuum aspiration are randomised to receive music therapy during the procedure.
  Interventions: Behavioral: music therapy
- Control (No Intervention): Routine Care

INTERVENTIONS:
Behavioral: music therapy — cases will randomly assigned to receive music therapy group with routine care, plus music given via headphone, or assign to control group with no music given.
  Other Names: No music therapy; Routine Care
  Arms: MVA case undergone music therapy

SUMMARY:
Manual vacuum aspiration (MVA) is one of the surgical treatment options for managing early pregnancy loss. When compared to traditional surgical method; MVA is safer, more cost-effective, due to its shorter hospitalisation period and not undergo the risk of general anaesthesia. The MVA procedure is performed under local anaesthesia and analgesics is given prior the procedure. However, majority of patients still complaint significant pain during the procedure.

In our previous study, the investigator found women had high anxiety and stress levels when undergo miscarriage and the operation. Pain perception may further be affected by one's psychological state at the time of the procedure. Therefore reducing the patient's anxiety during the USG-MVA may further improve the patient's pain control and overall acceptance of the procedure.

Music can act as a distracter and has a calming effect which turn the patient's attention away from negative stimuli. Yet, there has been no RCTs to investigate the beneficial effect of music therapy in pain control or reducing anxiety levels during USG-MVA.

The investigator hypothesis the intervention of music therapy to our current pain control will reduce the pain and anxiety levels experienced by our patients during USG-MVA. Thus, there is a need to conduct an RCT to test our hypothesis.

The study is conducted in an university affilated hospital for women undergo the USG-MVA procedure. The primary outcome is to evaluate in between group difference in the pain intensity after the USG-guided MVA procedure. The secondary outcome is to evaluate the difference in anxiety level . Case is randomized to music and non music group, Bluetooth headphone are provided during the procedure and case can choose their favourite songs. The outcome are measured by the self rated instrument: Visual analogue scale and the STAI trait anxiety score and the physiological measure salivary alpha amylase (sAA )score. The pain score and the anxiety level is measured pre operatively, immediate after the procedure and 2 hours post operatively. The SPSS-26 will be used for statistics analysis.

DETAILED DESCRIPTION:
Title: The efficacy of music as an adjunct analgesic in reducing pain and anxiety during ultrasound-guided manual vacuum aspiration (USG-MVA): A randomized controlled trial.

Approximately one in four women will experience an early pregnancy loss in her lifetime. Manual vacuum aspiration (MVA) is one of the treatment options for managing early pregnancy loss. USG-MVA is safer, more cost-effective, and is associated with shorter hospital stay and cost than traditional surgical method. However, majority of patients experience significant pain during the procedure.

At present, there is no consensus on the optimal pain control regimen for USG-MVA. The pain generated from USG-MVA may be due to the dilatation of the cervix or insertion of the catheter or due to uterine contraction. Various analgesic methods have been used to reduce the pain including the use of paracervical block (PCB), non-steroidal anti-inflammatory drugs (NSAIDs), lidocaine gel and conscious sedation but the procedure is still not absolutely painless. Pain management remains an important factor in its success and patient acceptance.

In our previous study, the investigator evaluated the effectiveness of adding Buscopan®, an anti-spasmodic agent, as pain control regimen for women undergone the USG-MVA. Result found that the intervention group were more satisfied to the procedure than the placebo group. They had 15% and 21% lower pain score immediately after the operation as well as two hours post operatively. The investigator postulated the women receiving Buscopan® is being relieved from experiencing uterine spasms. However, the investigator found that the women had higher anxiety levels as reflected by the high anxiety scores in their Hospital Anxiety Depression Scale. Pain perception maybe affected by one's psychological state at the time of the procedure. And undergo a surgical procedure plus the diagnosis of miscarriage further increases their anxiety and stress levels. Therefore to reduce the patient's anxiety during the USG-MVA may further improve the patient's pain control and overall acceptance of the procedure.

Music is known to have a calming effect; previous studies have postulated that music can act as a distracter which turns the patient's attention away from negative stimuli. Another theory is that music activates brain as rewarding region which is responsible for pleasant experiences and happiness and induces dopamine release in striatal system. A systematic review of 42 randomized controlled trials of music interventions in the preoperative setting found music significantly reduced anxiety and pain. Previous studies also showed music as an auxiliary analgesic during first trimester surgical abortion but only with small sample size and mixed results. There has not been any RCTs to investigate the beneficial effect of music therapy in pain control or reducing anxiety levels during USG-MVA.

we hypothesis the addition of music to our current pain control can reduce pain and anxiety levels experienced by our patients during USG-MVA.

The Primary outcome is to evaluate the difference in pain score immediate postoperative and 2 hours after the USG-guided MVA procedure between the intervention and control groups. The Secondary outcome is to evaluate the difference in their anxiety levels.

Plan of Investigation:

Subjects All women undergoing USG- MVA for the treatment of early pregnancy loss with gestation less than 12 weeks; size of the gestation product is less than 5 cm.

Inclusion criteria includes:

Women 18 years old or above Women with miscarriage who are feasible for USG-MVA

Exclusion criteria includes:

Not feasible for MVA procedure Partial or total hearing impairment on analgesic or anxiolytic before admission to hospital. Patient refusal

(ii) Methods The patient is recruited in the Department of Obstetrics and Gynaecology in a university base hospital. The participates consented for the USG-MVA procedure.

Randomization For those who consented to the study, they will randomly assign to receive music therapy or not, according to a computer generated random number series in 1:1 ratio. Each number will be placed in an opaque envelope labelled serially: (i) intervention group: routine USG-MVA procedure plus music given via headphone (ii) control group- routine USG-MVA procedure with no music given, with no headphone is given either. Given the audible and physical features of the intervention, it is impossible to blind the participant and physicians, staff and research assistant in the process.

USG-MVA procedure (Routine care)

USG-MVA will carry out in an outpatient day ward. Women will be given oral Misoprostol tablet 2-3 hours before the procedure for cervical priming. All patients will be given naproxen (500 mg) orally an hour and an intravenous injection of Buscopan® (20mg) 5 minutes before the procedure. If the woman is allergic to NSAIDs, paracetamol or codeine will be used instead. The women will be asked to have full bladder for the abdominal USG.

During the USG-MVA procedure, the women are placed in the lithotomy position and aseptically dressed. Speculum will be put to visualize the cervix. 5 ml 2% xylocaine local anaesthetic will be injected at the cervical-vaginal juncture at 4, 5,7, 8 o'clock position. The anterior lip of cervix is held with a volsellum and cervical dilation is performed if required. A 60ml charged syringe will attach to the curette (size 4 to 7mm). 5ml 2% Xylocaine gel will be applied to the cervical canal and over the end of the curette tip during the insertion. And abdominal USG will be performed during the procedure to ensure complete evacuation and prevent perforation of organs.

The USG-MVA will stop as soon as USG confirm that the uterine cavity was empty. Any post-operative complications including significant bleeding requiring blood transfusion, uterine perforation and infection will be recorded. Women will be discharged after two hours if they were stable. And they are asked to return 3 weeks later for a pregnancy test to evaluate the completeness of evacuation.

Intervention group (Music therapy)

In additional to the standard routine care, the patients are asked to select their favourite music; they will start to hear the music when they are placed in lithotomy position and end when procedure completed (removal speculum). They are asked not to hear any music before and after the procedure. A bluetooth headphone fitted with sanitary covers is offered. The volume of the media player is preset so instructions from the staff or clinicians could still be heard. The genre of music chosen will be recorded.

Control group (No Music) In the control group, neither music nor headphones will be offered. The participants are also asked not to listen to any music before; during or after the USG-MVA and they will undergo the routine USG-MVA procedure.

Pain assessment Participants are asked to rate their pain intensity by the visual analog scale (VAS). The scores ranged from 0 to 100, where 0 indicated no pain and 100 indicated the worst pain imaginable. The pain score will be assessed when participants enter the department, 30 minutes after administration of misoprostol, at the end of the procedure and 2 hours after the procedure. The need for additional postoperative analgesics were recorded (yes or no).

Stress and Anxiety levels The participants anxiety and stress level are assessed by the Chinese version of the General Health Questionnaire-12 (GHQ-12), Hospital Anxiety and Depression Scale (HADS) and State anxiety (STAI-S) of the State-trait Anxiety Inventory and the salivary alpha amylase level.

General health questionnaire (GHQ-12) The participants preoperative anxiety level are assessed by the GHQ-12. It consists a 4-point Likert ranging from 1 to 4; The total score ranges from 12-48, score greater than 27 indicate a higher level of psychological distress.

Hospital Anxiety and Depression Scale (HADS) The HADS aims to evaluate the participants their state of anxiety and depression. It is a 4-point Likert ranging from 0 to 3. The total score ranges from 0 to 21. The cut-off point is 8 for higher state of anxiety or depression.

State-trait anxiety inventory- State Anxiety Subscale (STAI-S) The STAI-S aims to evaluate the current state of anxiety. Participants are asked to answer the questionnaires during admission, after 30 minutes of cytotec administration, immediate and 2 hours after the USG-MVA. It consists of 20 questions with 4 points Likert scale. The total scores range from 20 to 80, with higher scores correlating with greater anxiety.

Stress biomarker assessment -Salivary alpha amylase (SAA) The Salivary alpha-amylase (sAA) levels measures the physiological stress, they are collected by a dedicated SaliCap® collection device via the passive drooling method before; immediately and at 30 minutes after MVA procedure. All patients were asked not to eat or drink at least an hour before collection.

Client satisfaction assessment

Client Satisfaction Questionnaire (CSQ) It is a self-administered questionnaire to assess client satisfaction and acceptance. It consists of eight items with 4-point Likert Scale, from "Very satisfied" to "Quite dissatisfied".

(iv) Data processing and analysis Statistical Analysis All statistical analyses will be performed using SPSS 22.0 based on intention-to-treat. A two-tailed probability value of p< 0.05 will be considered statistically significant.

Sample size Previous studies in women undergoing gynaecological procedures reported that music therapy could reduce pain scores by between 35% to 50%. Assuming an alpha of 0.05, power of 90% , estimated that 73 participants will be recruited in each group to detect a 1- sided medium effect size of 0.5 due to music therapy. To allow for 20% drop-out rate, the planned sample size will be increased to 88 per group.

Duration of study Aim to conduct for 18 months, followed by 6 months for data collection and analysis. Patients' recruitment will start after ethics approval.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or above
* hospitalized for termination of first trimester pregnancy under local anaesthesia

Exclusion Criteria:

* being a minor or adult protected by law
* not feasible for MVA procedure
* Partial or total hearing impairment
* on anxiolytics and analgesics before arriving at the hospital
* refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — First trimester miscarriage women.
Enrollment: 176 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
To assess the change in post operatively pain score with or without MT at different time points | During one day
  The case self rated the VAS score, VAS scores ranged from 0 to 100, where 0 indicated no pain and 100 indicated the worst pain imaginable.
  (T0) when entering the department, (T1) 30 minutes after administration of misoprostol, (T2) during the procedure, (T3) at the end of the procedure and (T4) 2 hours after the procedure.

SECONDARY OUTCOMES:
To assess the impact of MT on anxiety level | During one day
  The client self rated the Chinese version of STAI-S subscore. It is a 20 item scale with a 4 point likert ranging from almost never to almost always. the total scores range from 20 to 80, with higher scores correlate with greater anxiety.
To assess the psychological distress during the past few weeks | 1 hour before the procedure
  The client self rated the Chinese version General Health Questionnaire, it consists of 12 questions with 4 likert point rating. It aims to evaluate whether there are any baseline psychological distress, higher score indicates a higher level of psychological morbidity.
To assess the patient's satisfaction and acceptance | 2 hours after the procedure
  The client self rated the Client Satisfaction Questionnaire, it consists of 12 questions with 4 likert point rating. Higher score indicates greater acceptance and satisfaction
To measure the patient's physiological stress level. | Saliva samples were collected 1 hour before the procedure and 30 minutes after MVA procedure
  Saliva samples were collected via the passive drooling method , using a dedicated SaliCap collection device. All patients were asked not to eat or drink 1 hour before collection. The level is determined using the Indiko (Thermo Fisher Scientific) random access analyser to measure the physiological stress.

OTHER OUTCOMES:
To assess any post operative physical discomfort | immediate after post operative and 2 hours post operatively
  The case will complete the questionnaire of 4-likert point, with no, mild, moderate and severe for symptoms of nausea, vomiting, dizziness, tiredness, shortness of breath

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah Jacqueline Chung, MBBS, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No